CLINICAL TRIAL: NCT06348758
Title: Knowledge, Attitudes, And Perceptions of a Group of Egyptian Dental Students Towards Artificial Intelligence: A Cross-sectional Study
Brief Title: Knowledge, Attitudes, And Perceptions of a Group of Egyptian Dental Students Towards Artificial Intelligence
Acronym: AIKnowledge
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Fouad Wahby, Lecturer, Cairo University
Other Study IDs: KAP towards AI
Record Dates: First submitted 2024-03-14; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental Students in Egyptian Dental schools: Students should be in Egyptian Dental faculties. 1st year students will be excluded
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — E-Questionnaire will be sent to the students

SUMMARY:
In the context of this ongoing AI revolution, it is essential to ensure that current and future clinical practitioners are up to date regarding this technology's current state and potential. It is valuable to assess the current attitude of clinical dentists and undergraduate students in dentistry regarding the future role of AI.

To the best of the author's knowledge, there is no study about Egyptian dental students' views and attitudes regarding the application of AI in dental practice. Therefore, this study aimed to evaluate the attitudes and perceptions of a group of dental students in Egypt towards AI.

DETAILED DESCRIPTION:
Data will be collected using a questionnaire. The survey will be distributed to dental students at the Faculty of Dentistry, Cairo, and Egyptian Russian universities through Google Forms. The questionnaire comprised 3 sections and 22 questions. The survey consisted of a question on demographics and educational information about dental students, knowledge of and attitudes towards AI, future application areas of AI in dentistry, and topics of AI in dental education. The first part of the survey. Informed consent will be obtained from all the participants before completing the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Dental students

Exclusion Criteria:

* Graduates

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Dental students in Egypt
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-08-07 (Estimated)

PRIMARY OUTCOMES:
knowledge, attitudes, and perceptions about artificial intelligence in Dentistry | up to 6 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reem Wahby, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo University- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The results of the survey will be published after statistical analysis
Supporting Information: SAP
Time Frame: 1 year
Access Criteria: not available yet

REFERENCES:
- [Derived] Elchaghaby M, Wahby R. Knowledge, attitudes, and perceptions of a group of Egyptian dental students toward artificial intelligence: a cross-sectional study. BMC Oral Health. 2025 Jan 3;25(1):11. doi: 10.1186/s12903-024-05282-7. PMID 39754101